CLINICAL TRIAL: NCT04783272
Title: Photoacoustic Computed Tomography for Pre-Operative Reconstructive Flap Angiography - Pilot Study
Brief Title: Photoacoustic Computed Tomography for Pre-Operative Reconstructive Flap Angiography
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to use equipment at partner institution.
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Edward Ray, Principal Investigator, MD, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000648
Record Dates: First submitted 2021-02-17; First posted 2021-03-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Other Reconstructive Surgery; Plastic Surgery
Keywords: flap reconstructive surgery; Plastic Surgery; Photoacoustic Computed Tomography (PACT)
MeSH Terms: interventions — Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Treatment (Experimental): Photoacoustic Computed Tomography (PACT) Imaging
  Interventions: Diagnostic Test: Photoacoustic Computed Tomography (PACT) Imaging

INTERVENTIONS:
Diagnostic Test: Photoacoustic Computed Tomography (PACT) Imaging — PACT will be completed prior surgery.

SUMMARY:
The purpose of this study is to determine if a new non-invasive imaging technology, called Photoacoustic Computed Tomography (PACT), can be used in the pre-operative setting to better visualize the blood supply of reconstructive flaps used in Plastic Surgery.

DETAILED DESCRIPTION:
Photoacoustic Computed Tomography (PACT) is a novel, non-invasive imaging technique which can perform deep tissue imaging with high spatial resolution and optical contrast. The system utilizes short-pulsed lasers to generate photoacoustic waves in biological tissues. These are then detected by a 512-element full-ring transducer array, which allows for high spatial resolution, especially in deep tissues. In addition, PACT utilizes diffuse optical tomography, in which the light absorption of hemoglobin at visible or near-infrared wavelengths, provides excellent contrast for the imaging of human vasculature.

Prior studies of PACT imaging have evaluated this technique to image the human breast as an alternative modality for breast cancer screening as well as to image human extremities for the evaluation of vascular disease. The full-ring transducer array offers a significant advantage in spatial resolution, especially in deep tissues, over the standard linear arrays employed in the standard, widely-used handheld ultrasonic transducers. In addition, diffuse optical tomography allows for strong vascular contrast over a large field of view without the use of exogenous contrast agents.

Flap reconstructive surgery utilizes a patient's own soft tissues to recreate structures, fill large soft tissue defects, provide joint coverage, or perform other reconstructive operations. Examples of patients who would require flap reconstructive surgery include patients undergoing mastectomies and patients who have suffered from trauma with significant tissue loss. Tissue flaps have a defined blood supply which originate from the original site of the tissue. The flap can be compromised if the arterial supply or venous drainage is jeopardized during tissue transfer. Therefore, an accurate understanding of the blood supply of the tissue flap is crucial for successful flap reconstructive surgery.

Current pre-operative vascular imaging modalities for flap reconstructive surgery include handheld Doppler ultrasonography, magnetic resonance angiography (MRA), and the gold standard computed tomography angiography (CTA). Doppler ultrasonography is technician-dependent, inaccurate, and lacks optical contrast. MRA is expensive, requires a lengthy imaging time, and requires the administration of intravenous contrast. CTA is also expensive, also requires the administration of intravenous contrast, and requires the administration of ionizing radiation. PACT does not require the administration of intravenous contrast or ionizing radiation, and provides excellent spatial resolution and optical contrast. Therefore, PACT would be an optimal pre-operative vascular imaging modality for flap reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 who are planned to undergo non-urgent flap reconstructive surgery, specifically either an abdominally-based flap or an ALT flap, will be study candidates.

Exclusion Criteria:

* Patients who require urgent or emergent flap reconstructive surgery, have undergone prior abdominally-based or ALT flap reconstructive surgery, who cannot receive ionizing radiation (required for CTA), who cannot receive iodinated intravenous contrast (required for CTA), and whose weight exceeds 300lbs (weight limit of PACT machine) will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
PACT Patient Comfort Questionnaire | This questionnaire will be completed by patient at the time of the PACT Imaging visit. Imaging visit will occur after the initial visit and before surgery up to 4 months.
  The data is ordinal and discrete (Likert scale). The scale is 1 to 5 where 1 is the worst and 5 is the best.
Vascular Imaging Modality for Flap Reconstructive Surgery Questionnaire | This questionnaire will be completed by Dr. Edward Ray immediately following surgery.
  The data is ordinal and discrete (Likert scale). The scale is 1 to 5 where 1 is the worst and 5 is the best.

CONTACTS AND LOCATIONS:
Overall Officials: Edward Ray, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States